CLINICAL TRIAL: NCT01345877
Title: Pain Sensitivity in Acute Inflammatory Pain - Gender Differences and Validity of Sensory Tests
Brief Title: Pain Sensitivity in Acute Inflammatory Pain
Acronym: PASORI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Norpharma A/S (Industry)
Responsible Party: Principal Investigator, mads u werner, MD, DMSci, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-1-2009-132
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteers Are Studied
Keywords: burn injury; cold pressor test; gender; pain; pain sensitivity; pain prediction; psychometrics; quantitative sensory testing
MeSH Terms: conditions — Burns; Coitus; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gender (Other)
  Interventions: Procedure: first degree cutaneous burn injury

INTERVENTIONS:
Procedure: first degree cutaneous burn injury — application of thermode (5 x 2.5 cm) to lower leg temperature 47.0 C, 420 s
  Other Names: Modular Sensory Analyzer Thermotest (Somedic, Hörby, Sweden)

SUMMARY:
Pain is a complex experience influenced by gender and genetics, and, by psychosocial and sensory experiences. Pain sensitivity is thus highly variable between individuals.

In the present study we evaluate individuals´ pain perception in response to a number of different pain stimuli in 100 healthy volunteers (50 females and 50 males).

The data will allow us to assess pain sensitivity, to predict pain responses and to investigate gender related differences in pain perception.

A second aim is to evaluate the robustness of the different pain-tests since the tests are repeated with an interval of 2-4 weeks.

DETAILED DESCRIPTION:
Pain perception is affected by physiological, psychological, existential and demographic factors.

In the present study psychophysiological, psychological, genetic and demographic components in pain perception are evaluated in healthy volunteers (n = 100).

Psychophysical assessments following induction of a first degree burn injury (47.0 C, 420 s, 12.5 sq.cm, lower leg) include:

* pain during induction of burn injury
* thermal thresholds
* tactile thresholds
* electrical thresholds
* areas of secondary hyperalgesia
* pressure algometric assessments
* assessment of Diffuse Noxious Inhibitory Control (DNIC) efficiency
* assessment of (DNIC) using cold pressor test

Psychological assessments include:

* HADS (Hospital Anxiety and Depression Scale)
* PCS (Pain Catastrophizing Scale)
* vulnerability score

Genetics include:

- A118G SNP

Demographics include:

* gender
* height
* weight

ELIGIBILITY:
Inclusion Criteria:

* healthy
* psychomotor ability to perform the tests
* cognitive ability to perform the tests

Exclusion Criteria:

* smoker
* Body Mass Index > 28
* participation in drug studies < 4 weeks prior to inclusion
* chronic pain
* chronic intake of analgesics
* drug or alcohol abuse
* intake of analgesics < 48 hours prior to study
* females not on contraceptive therapy (intra-uterine device or p-pill)
* lesion in the assessment area

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
pain following burn injury | from baseline to 420 s after burn injury

SECONDARY OUTCOMES:
thermal thresholds | followed for 180 min after burn injury
tactile thresholds | followed for 180 min after burn injury
pressure algometry assessments | 95 min prior to burn injury
DNIC-efficiency | 45 min before burn injury
cold pressor test | 85 min before burn injury
HADS score | 2 hours before the burn injury
PCS ratings | 2 hours before the burn injury
A118G SNP | 8 months after inclusion completed

CONTACTS AND LOCATIONS:
Overall Officials: Mads U Werner, MD, DMSc, Principal Investigator — Multidsciplinary Pain Center 7612, Neuroscience Center, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Multidisciplinary Pain Center 7612, Neuroscience Center, Rigshospitalet, Blegdamsvej 9, Copenhagen O, Denmark

REFERENCES:
- [Background] Luginbuhl M, Schnider TW, Petersen-Felix S, Arendt-Nielsen L, Zbinden AM. Comparison of five experimental pain tests to measure analgesic effects of alfentanil. Anesthesiology. 2001 Jul;95(1):22-9. doi: 10.1097/00000542-200107000-00009. PMID 11465562
- [Background] Edwards RR, Fillingim RB, Ness TJ. Age-related differences in endogenous pain modulation: a comparison of diffuse noxious inhibitory controls in healthy older and younger adults. Pain. 2003 Jan;101(1-2):155-65. doi: 10.1016/s0304-3959(02)00324-x. PMID 12507710
- [Background] Neziri AY, Scaramozzino P, Andersen OK, Dickenson AH, Arendt-Nielsen L, Curatolo M. Reference values of mechanical and thermal pain tests in a pain-free population. Eur J Pain. 2011 Apr;15(4):376-83. doi: 10.1016/j.ejpain.2010.08.011. Epub 2010 Oct 6. PMID 20932788
- [Background] Neziri AY, Curatolo M, Nuesch E, Scaramozzino P, Andersen OK, Arendt-Nielsen L, Juni P. Factor analysis of responses to thermal, electrical, and mechanical painful stimuli supports the importance of multi-modal pain assessment. Pain. 2011 May;152(5):1146-1155. doi: 10.1016/j.pain.2011.01.047. Epub 2011 Mar 10. PMID 21396782
- [Result] Ravn P, Frederiksen R, Skovsen AP, Christrup LL, Werner MU. Prediction of pain sensitivity in healthy volunteers. J Pain Res. 2012;5:313-26. doi: 10.2147/JPR.S33925. Epub 2012 Aug 29. PMID 23055774